CLINICAL TRIAL: NCT01408537
Title: Immunogenicity and Safety of Inactivated Vero Cell Derived Japanese Encephalitis Vaccine in Thai Children
Acronym: JE0153
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Pornthep Chanthavanich, Department of Tropical Pediatrics, Faculty of Tropical Medicine, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JE0153
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Encephalitis, Japanese B
Keywords: inactivated Japanese encephalitis vaccine; vero cell; children; immunogenicity; safety
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JEVAC (Experimental): JEVAC 0.5 mL/ dose subcutaneously injected on upper thigh at D0, 1-4wk, and 1 year
  Interventions: Biological: JEVAC

INTERVENTIONS:
Biological: JEVAC — Each subject will receive 3 doses of JEVAC subcutaneously on Day 0, 1-4 weeks and a booster vaccination at one year. Each dose of JEVAC contains 0.5 mL. of inactivated Vero cell derived JE vaccine (Beijing P-3 strain).

SUMMARY:
Japanese encephalitis (JE) is the main cause of viral encephalitis in many countries of Asia including Thailand. Estimated annual mortality ranges from10,000-15,000 deaths, while the total number of clinical cases is about 50,000. Of these cases, about 50% result in permanent neuropsychiatric sequelae. The disease occurs mostly among children aged <10 years. There is no specific antiviral treatment for JE. Vaccination is the single most important control measure. This study aims to evaluate the immunogenicity and safety of inactivated Vero cell derived JE vaccine (Beijing P-3 strain) produced by Liaoning Cheng Da Biotechnology Co., Ltd, China "JEVAC" in Thai children.

152 healthy Thai children aged between 1-3 years will be vaccinated with "JEVAC" in a dose of 0.5 mL. subcutaneously on Day 0, 1-4 weeks later and a booster vaccination at one year (totally 3 doses). Two mL. of blood will be drawn on Day 0, 4 weeks after second dose, at one year on booster vaccination day and 4 weeks after the booster (totally 8 mL. of 13 months study period) for determination of JE neutralizing antibodies (PRNT50) using Beijing P3 strain. Adverse events will be observed for 28 days after each vaccination. Serious adverse events will be observed throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Thai children aged 1- 3 years
2. No previous history of JE vaccination
3. Available for all visited schedule in the study period.
4. Written inform consent signed by a parent or guardian

Exclusion Criteria:

1. Known serious underlying diseases such as nervous system, heart, kidney and liver diseases.
2. Known hypersensitivity to JE vaccine composition such as human albumin, dextran 40, etc.
3. Previous history of JE disease.
4. Receive the blood component within the past 3 months,
5. Known history of immunocompromised conditions such as HIV/AIDS, malignancy.
6. Under treatment of immunosuppressive drugs such as systemic corticosteroid and anti-neoplastic drug.
7. Febrile illness (temperature ≥37.5°C) or acute illness/infection on the day of vaccination
8. Plan to leave the study area before the end of study period.
9. Participating in other clinical trials.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2010-05; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pornthep Chanthavanich, MD, Principal Investigator — Department of Tropical Pediatrics, Faculty of Tropical Medicine, Mahidol University
Locations (1):
- Department Tropical Pediatrics, Ratchathewi, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment took place in 2 sites (Department of Tropical Pediatrics, Faculty of Tropical Medicine and Nopparat Rajathanee Hospital) from 3rd May 2010 to 10th August 2010. One hundred and fifty two subjects who illegible for the inclusion and exclusion criteria were enrolled in the study.
Pre-assignment Details: There was no subject who did not get the study vaccine after informed consent was signed.
Groups:
- JEVAC: JEVAC : Each subject will receive 3 doses of JEVAC subcutaneously on Day 0, 1-4 weeks and a booster vaccination at one year. Each dose of JEVAC contains 0.5 mL. of inactivated Vero cell derived JE vaccine (Beijing P-3 strain).
Period: Overall Study
Arm/Group | JEVAC
Started | 152
Completed | 144
Not Completed | 8
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | JEVAC
Number analyzed (Participants) | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 152
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.2 (0.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 79

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion Rate After Primary Vaccination
Description: To determine the seroconversion rate by using neutralizing antibody (NT) against JE virus (Beijing P3 strain) JE virus from <10 on before first vaccination To >= 10 at 28 days after second vaccination (primary vaccination). Those who have NT titer >=10 before first vaccination, will not be included in immunogenicity evaluation.
Time Frame: 28 days after second dose of JEVAC
Population: There were 152 enrolled subjects in the study. However, 5 subjects had NT titer >= 10 before first vaccination and one subject whom blood on 28days after second vaccination was not drawn due to withdrawn consent. Therefore, the number of subjects for the outcome measurement should be 146.
Measure: Number; unit: percentage of seroconversion
Arm/Group | JEVAC
Number analyzed (Participants) | 146
percentage of seroconversion | 100

2. Secondary Outcome: Geometric Mean Titer of NT After Primary and Booster Vaccination
Description: To determine the geometric mean titers (GMT) of neutralizing antibody of JEVAC 1 month after primary and then before and after booster vaccinations.
Time Frame: 28 days after second vaccination, before and 28 days after booster vaccination with JEVAC
Population: 152 were enrolled, 1 withdrawn consent before second vaccine, 5 had NT >= 10 before first vaccine, 146 included in D28 after second vaccine. At 1 year, 3 received JE vaccine outside the study, 3 lost follow up, 140 included in before booster, At D28 after booster, 1 could not draw blood, 139 included in D28 after booster.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- GMT of NT on 28days After Vaccination: GMT of NT titer of subjects on 28 days after vaccination (excluded the subject who had NT titer > =10 before first vaccination).
- GMT of NT Before Booster Vaccine: GMT of NT of subject at 1 year before booster vaccination. Exclude NT titer >=10 before first vaccination and subjects received JE vaccine outside the study.
- GMT of NT Titer After Booster Vaccine: GMT of NT of subject at 28 days after booster vaccination. Exclude NT titer >=10 before first vaccination and subjects received JE vaccine outside the study.
Arm/Group | GMT of NT on 28days After Vaccination | GMT of NT Before Booster Vaccine | GMT of NT Titer After Booster Vaccine
Number analyzed (Participants) | 146 | 140 | 139
titer | 150.01 [126.4 to 175.7] | 49.33 [39.0 to 62.4] | 621.66 [510.4 to 757.2]

3. Secondary Outcome: Adverse Events of Vaccine
Description: To determine the adverse events of JEVAC
Time Frame: 7, 14, 28 days after each vaccination and throughout the study period for local, solicited systemic, unsolicited systemic and serious adverse events, respectively
Population: Determined AEs by number of injections 152 injection for the first dose 151 injection for the second dose 145 injection for the third dose
Measure: Number; unit: events
Units Other Than Participants: injections
Groups:
- Fever After Vaccination: Fever (Temp > =37.5 Axillary )after each vaccinations (3 doses). Episode of fever was collected up to 28 days after each vaccination.
- Local AE JEVAC After Vaccination: Local Adverse event (tenderness, redness, ecchymosis, hematoma and swelling) after each vaccinations the first vaccination was on day of enrollment, the second dose was Day7 (+21day))
  , Booster vaccine was on 1 year(+30days). Local AEs were collected up to 28 days after each vaccination.
- Chills After Vaccination: Chills after each vaccinations (3 doses). Episode of chills was collected up to 28 days after each vaccination.
- Poor Appetite After Vaccination: Poor appetite after each vaccinations (3 doses). Episode of poor appetite was collected up to 28 days after each vaccination.
- Vomiting After Vaccination: Vomiting after each vaccinations (3 doses). Episode of vomiting was collected up to 28 days after each vaccination.
- Urticaria After Vaccination: Urticaria after each vaccinations (3 doses). Episode of Urticaria was collected up to 28 days after each vaccination.
- Unsolicited AEs After Each Vaccination: unsolicited AEs after each vaccinations (3 doses). Episode of unsolicited AEs (excluded SAEs) were collected up to 28 days after each vaccination
- SAEs Entire the Study: SAEs which occured entire the study period were recorded.
Arm/Group | Fever After Vaccination | Local AE JEVAC After Vaccination | Chills After Vaccination | Poor Appetite After Vaccination | Vomiting After Vaccination | Urticaria After Vaccination | Unsolicited AEs After Each Vaccination | SAEs Entire the Study
Number analyzed (Participants) | 152 | 152 | 152 | 152 | 152 | 152 | 152 | 152
Number analyzed (injections) | 448 | 448 | 448 | 448 | 448 | 448 | 448 | 448
events | 79 | 5 | 3 | 24 | 36 | 3 | 63 | 21

4. Secondary Outcome: Neutralizing Antibody Persistence One Year After the Primary Vaccination
Description: To determine the neutralizing antibody persistence one year after the primary JEVAC vaccination.
Time Frame: 1 year after primary vaccination
Population: The analysis was excluded 5 subjects who had NT titer >10 on D0
Measure: Number; unit: participants
Arm/Group | JEVAC
Number analyzed (Participants) | 140
participants | 125

ADVERSE EVENTS:
Time Frame: In addition to systematic assessment on Day 0-14 after each vaccination, Any unsolicited AE was accessed within 28 days after each vaccination. Any SAE was accessed through the study period (1 yr +28 days).
Arm/Group | JEVAC
Serious Adverse Events (participants affected / at risk) | 21/152
Other Adverse Events (participants affected / at risk) | 89/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JEVAC (N=152)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 (6)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 4 (4)
skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
seizure (Nervous system disorders) | 5 (5)
infection (other) (Infections and infestations) | 2 (2)
pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JEVAC (N=152)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 27 (27)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
diarrhea (Gastrointestinal disorders) | 9 (9)
vomiting (Gastrointestinal disorders) | 1 (1)
skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
infection (Infections and infestations) | 7 (7)
contact dermatitis (Skin and subcutaneous tissue disorders) | 13 (13)
Fever (Infections and infestations) | 64 (79) — Axillary temperature greater than or equal 37.5 celsius
chills (Infections and infestations) | 3 (3)
poor appetite (Gastrointestinal disorders) | 22 (24)
vomiting (Gastrointestinal disorders) | 32 (36)
urticaria (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No